CLINICAL TRIAL: NCT05551650
Title: Early Life Social, Environmental, and Nutritional Determinants of Disease
Brief Title: El Sendero: Pathways to Health Study
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: University of Colorado, Denver (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Michael I. Goran, Principal Investigator, University of Southern California
Other Study IDs: CHLA-21-00314
Record Dates: First submitted 2022-08-08; First posted 2022-09-23 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Obesity, Childhood; Child Development
Keywords: Childhood; Brain development; Adiposity; Nutrition; HMOs; Air-pollution
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project will continue to follow two birth cohorts of mother-infant Latino dyads through a series of new assessments at age 6y, with an emphasis on examining the the role early nutritional exposures, exposures to environmental toxins, and social determinants of health have on adiposity, eating behaviors, brain structure and function, cognitive outcomes, and chronic disease risk.

DETAILED DESCRIPTION:
This project will continue our work in two birth cohorts of mother-infant Latino dyads (NCT04434027 & NCT03141346) through a series of new assessments at age 6y, with a focus on examining the role of early nutritional exposures, exposures to environmental toxins, and social determinants of health (SDOH) on adiposity, eating behaviors, brain structure and function, cognitive outcomes, and chronic disease risk. This collection of assessments at 6 years of age is funded by two grants (R01 DK110793 01A1 & P50 MD017344). Breast milk has been shown to contain certain macronutrients (human milk oligosaccharides; HMOs) that vary greatly among women. Research from our lab recently characterized associations of HMOs with infant obesity, eating behaviors, and brain development as well as dynamic changes in HMOs over the course of breastfeeding and suggests that these factors are significant predictors of infant weight gain and adiposity. Additionally, we already obtained detailed individual measures of ambient and near-roadway air pollution exposure from pregnancy to 2y of age. Our previous work in a subset of participants from the proposed cohort found that increased prenatal exposure to ambient air pollutants was associated with increased infant growth and adiposity after adjusting for infant sex and age, pre-pregnancy BMI, breastfeeding, maternal age, season of birth, and SES. By conducting longer-term follow-up with more rigorous outcomes at age 6y, we will be able to more definitively determine if and how early nutrition, particularly specific HMOs, impact chronic disease risk in Latino children as well as how environmental exposure to toxins and the food environment may exacerbate these health outcomes. Here, we will explore:

1. The impact of infant exposure to environmental toxins on subclinical markers of chronic disease risk at age 6y.
2. The impact of infant exposure to environmental toxins and nutrition, especially the HMOs 2'FL, LNFPI, LNFPII, LNnT & LNH, in early life on adiposity and chronic disease risk at age 6y.
3. The impact of infant exposure to HMOs containing fructose and sialic acid on brain development at age 6y using image-based measures of brain structure (anatomical MRI), function (resting state fMRI), blood flow (arterial spin labeling), myelination and tissue microstructure (diffusion tensor imaging) as well as cognitive outcomes.
4. The impact of breast feeding (at breast vs delivered via a bottle) and the changing HMO profile on eating in the absence of hunger at age 6y, and structural and functional differences in key areas of the brain involved with appetite regulation (frontal cortex, basal ganglia, hippocampus, hypothalamus).
5. The impact of the food environment and broader SDOH on subclinical markers of chronic disease and how these relationships may exacerbate the effects of poor nutrition and environmental toxins.

Exposures:

Ambient Air pollution: Addresses will be used to generate x,y coordinates of latitude and longitude, geoIDs, and census tracts. These spatial elements will be used to query several databases to generate new geocoded social and environmental exposure variables. In addition, child dates of birth will be used to assign air pollution exposure estimates and community contextual variables for relevant time windows in early life through 6 years of age. Ambient air pollution will be measured by assigning PM2.5, NO2, and O3 exposures using hybrid model outputs developed by a team lead by Dr. Joel Schwartz (Harvard) over many years.

Near-Roadway Air Pollution (NRAP) : Addresses will be used to generate x,y coordinates of latitude and longitude, geoIDs, and census tracts. These spatial elements will be used to query several databases to generate new geocoded social and environmental exposure variables. In addition, child dates of birth will be used to assign air pollution exposure estimates and community contextual variables for relevant time windows in early life through 6 years of age. NRAP is a complex mixture of particles and gases, including particulate matter, organic compounds, elemental carbon, and polycyclic aromatic hydrocarbons. In this study, NRAP exposure will be characterized using the CALINE4 air quality dispersion model that incorporate HERE (www.here.com) detailed roadway geometry, traffic volumes from Streetlytics™ by Citilabs, Inc. (www.citilabs.com), vehicle emission rates from CARB's EMFAC2017 model, and atmospheric transport and dispersion (using wind speed, wind direction, atmospheric stability, and height of the mixing layer).

Social Determinants of Health (SDH): Addresses will be used to generate x,y coordinates of latitude and longitude, geoIDs, and census tracts. These spatial elements will be used to query several databases to generate new geocoded social and environmental exposure variables. In addition, child dates of birth will be used to assign air pollution exposure estimates and community contextual variables for relevant time windows in early life through 6 years of age. To capture SHD, we will use both individual-level data obtained from self-reported instruments as well context-level data obtained through geocoding and enrichment of participant data. For our geospatial analysis, using patient home addresses, we will assign (x,y) geographical coordinates using GIS software, which are spatially joined or associated with census tract polygons into which they fall. An 11-digit "Spatial GeoID" is appended to each point. The GeoID is then used to match the relevant data point to data from several state and national databases, including the US Census Bureau, the American Communities Survey, the US Department of Agriculture Economic Research Service, the Environmental Protection Agency, the California Environmental Health Screen, and the Healthy Places Index. PhenX SDOH core constructs will be used to capture sex, marital status, household composition, race/ethnicity, age, gender identity, birthplace, English proficiency, health literacy employment, food insecurity, and access to health services. Maternal Social Health will be assessed using validated measures from the Patient-Reported Outcomes Measurement Information System (PROMIS®). Two key domains relevant to diet and chronic disease will be measured: social isolation and social support. Acculturation to the US will be assessed by the Marin Short Acculturation Scale.

Child Dietary Intake: 24-hour dietary and physical activity recalls will be conducted in triplicate (1 weekend day and 2 weekdays). Dietary intake will be analyzed using the most current version of NDSR, which has been used extensively in the Goran lab and elsewhere for studies in Hispanics. Diet will be assessed at 6y of age.

Child Physical Activity: To assess physical activity, we will use the early years physical activity questionnaire (EY-PAQ). Mothers will be asked to report the frequency and duration of different Moderate to vigorous physical activity and sedentary time in which their child engaged during a typical week in the previous month. Physical activity will be assessed at 6y of age.

Child Sleep: To assess sleep, we selected the Children's Sleep Habits Questionnaire172, because it captures all domains of sleep health and was designed for children aged 2-10 years. Child sleep will be assessed at 6y of age.

Previously collected exposures: Early nutrition including breastfeeding versus formula feeding, breastfeeding exclusivity, breastfeeding duration, Breastmilk composition including HMO concentrations, and dietary intake were assessed at the timepoints 1 month (baseline), 6 months, 12 months, 24 months and 36 months. All previously collected variables can be found at the ClinicalTrials.gov pages for the original two cohorts from which this project stems: The Effects of Natural Sugars in Breast Milk on Healthy Infant Growth and Development (NCT04434027) and Improving the Eating Habits of Mother and Her Infant Via Sugar Reduction (MAMITA) (NCT03141346).

ELIGIBILITY:
All participants will be recruited from two existing cohorts: The Effects of Natural Sugars in Breast Milk on Healthy Infant Growth and Development (NCT04434027) and Improving the Eating Habits of Mother and Her Infant Via Sugar Reduction (MAMITA) (NCT03141346). Children and their mother's will be eligible for this study at child 6 years of age.

Initial Inclusion Criteria:

* Mother's normal weight or overweight/obesity prior to pregnancy
* Mother's who self identify as Hispanic
* Mother's who are first-time moms
* Mother's who have or have had singleton births
* Mothers must be able/willing to understand the procedures of the study, and must be able to read English or Spanish at a 5th grade level

Initial Exclusion Criteria:

* Physician diagnosis of a major medical illness (including type 1 or type 2 diabetes) or eating disorder in mothers
* Physical, mental, or cognitive issues that prevent participation
* Chronic use of any medication that may affect body weight or composition, insulin resistance, or lipid profiles
* Current smoking (more than 1 cigarette in the past week) or use of other recreational drugs
* Clinical diagnosis of gestational diabetes
* Pre-term/low birth weight infants, or diagnosis of any fetal abnormalities
* Mothers less than 18 years of age at the time of delivery will not be eligible as to avoid potential confounding from those subjects who might still be completing adolescent growth

Ages: 6 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Normal, overweight or obese (>25 BMI kg/m2) non-diabetic Hispanic mothers (18-59yrs) and their children (6y) from Los Angeles, CA.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Child weight | 6 years old
  Weight (kg) will be measured using a portable digital scale.
Child height | 6 years old
  Height (cm) will be measured using a stadiometer.
Child BMI percentile at 6y | 6 years old
  Child height and weight will be used to calculate body mass index (BMI) and BMI percentiles.
Child abdominal fat mass as measured by MRI | 6 years old
  An abdominal MRI using a 3.0 Philips Achieva will be used to measure visceral versus subcutaneous abdominal fat, in grams.
Child Liver fat content as measured by MRI | 6 years old
  An abdominal MRI using a 3.0 Philips Achieva will be used to measure liver fat fraction, percent liver fat.
Child cognitive capacity | 6 years old
  The child's cognitive capacity will be measured using the NIH Toolbox Cognition Battery, which is a standardized psychometrically rigorous tablet-based testing of core neuropsychological functions. Cognitive assessments will focus on visual attention and inhibitory control, cognitive flexibility/concept formation, working memory capacity, episodic memory, information processing speed, vocabulary knowledge, and oral reading skills.
Child Brain imaging - Anatomical MRI | 6 years old
  A 3.0 Philips Achieva will be used to perform an anatomical MRI to measure the volume and shape of brain regions including thickness of the cortical mantle and local volumes (indentation and protrusions) of the cortical and white matter surfaces.
Child Brain imaging - Perfusion Imaging (ASL) | 6 years old
  A 3.0 Philips Achieva will be used to perform Perfusion Imaging (ASL) to quantify regional cerebral blood flow (rCBF) at rest.
Child Brain imaging - Resting-State Functional MRI (rs-fMRI) | 6 years old
  A 3.0 Philips Achieva will be used to perform a Resting-State Functional MRI (rs-fMRI) to measure correlations of neural activity between regions in the brain ("functional connectivity"). We will used Graph Theoretical Measures to characterize functional connectivity throughout the brain.
Child Brain imaging- Diffusion Tensor Imaging (DTI) | 6 years old
  A 3.0 Philips Achieva will be used to perform Diffusion Tensor Imaging (DTI) to assess tissue organization within the brain, especially white matter fibers that connect one brain region to another. Measures will include: Fractional Anisotropy (FA) measuring the directional diffusion of water; Mean Diffusivity (MD), measuring the overall diffusion of water; Axial Diffusivity (AD) and Radial Diffusivity (RD) will be used to measure diffusion along hte long axis of diffusion or perpendicular to it.

SECONDARY OUTCOMES:
Child feeding behavior | 6 years old
  The child eating behavior questionnaire (CEBQ) will be administered and completed by the child's mother at child age 6yr.
Child behavior -Temperament | 6 years old
  The Early Childhood Behavior Questionnaire will be administered and completed by the child's mother at child 6yr of age to assess temperament including "surgency/extraversion", "negative affectivity", and "effortful control".
Child glycemic control as measured by HbA1c | 6 years old
  HbA1c will be measured in a subset of children from fasting blood. Blood samples will be drawn using the Tasso OnDemand Blood collection kit.
Child glucose tolerance as measured by a continuous glucose monitor (CGM) | 6 years old
  A subset of children will wear a FreeStyle Libre Pro CGM for 7-14 days, which measures blood glucose every 15 minutes.
Child fasting lipid profile | 6 years old
  Lipids (total cholesterol, LDL, HDL) will be measured from fasting blood in a subset of children using the Tasso OnDemand Blood collection kit.
Child PNPLA3 genotyping | 6 years old
  High quality genomic DNA will be extracted from saliva using Oragene kits (OG-610) from Genotek. Genotyping for SNP rs738409 in PNPLA3 will be carried out using the restriction fragment length polymorphism analysis technique.
Child abdominal circumference | 6 years old
  Abdominal circumference will be measured at the umbilicus to the nearest 1 mm.
Child skinfold thickness | 6 years old
  Child skinfold thickness will be measured in duplicate using a commercial caliper at the following sites: tricep, subscapular, suprailiac, and midthigh.
Child gut microbiome composition | 6 years old
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Child fecal metabolomics | 6 years old
  Raw stool samples will be collected in ethanol and aliquoted to be stored at -80oC for future metabolomics analysis. We will utilize un-targeted metabolomic based on liquid chromatography (LC) with high-resolution metabolomics (HRM) to characterize endogenous and exogenous metabolites.
Child appetite regulation | 6 years old
  Child's appetite regulation will be measured through the eating in the absence of hunger (EAH) protocol. Briefly, after a standard meal, and assessment of level of fullness, child will have access to a variety of palatable, portioned, and weighed snack foods as well as a range of toys for a 10 minute free-access period. Pre- and post- weights of the snack foods will be used to determine the quantity of food consumed with higher energy consumption representing a higher degree of EAH.
Child non-verbal and fluid intelligence | 6 years old
  Nonverbal/fluid intelligence will be measured using the Raven's 2 Progressive Matrices test (short form), which provides a measure of intellectual capacity that minimizes the impacts of language skills and cultural differences.
Child mental and behavioral health- parent ratings | 6 years old
  Mothers will complete the Behavioral Assessment Scale for Children, 3rd ed (BASC-3).
Child executive function - parent ratings | 6 years old
  Mothers will complete the Behavior Rating iNventory of Executive Function (BRIEF).
Maternal weight | Child 6 years old
  Weight (kg) will be measured using a portable digital scale.
Maternal height | Child 6 years old
  Height (cm) will be measured using a stadiometer.
Maternal BMI | Child 6 years old
  Body Mass Index (BMI) will be calculated based on the equation (weight in kg)/(height in m)^2.
Maternal systolic and diastolic blood pressure at baseline | Child 6 years old
  Sitting systolic and diastolic blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States